CLINICAL TRIAL: NCT01574404
Title: Polar Body Biopsy (PB) for Preimplantation Genetic Screening
Brief Title: Polar Body Biopsy for Preimplantation Genetic Screening
Acronym: Polar Body
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0911010734
Record Dates: First submitted 2012-03-16; First posted 2012-04-10 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Aneuploidy
Keywords: PGS,PGD, IVF, Polar Body Biopsy, FISH, Microarray analysis
MeSH Terms: conditions — Aneuploidy | interventions — Phosphatidylglycerols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Polar Body Biopsy with PGS (Experimental): Polar Body Biopsy with Pre implantation genetic screening
  Interventions: Procedure: Polar body biopsy with PGS

INTERVENTIONS:
Procedure: Polar body biopsy with PGS — PB biopsy and analysis by comparing the PB results to the FISH/microarray results

SUMMARY:
People with infertility undergoing in vitro fertilization (IVF) can test the embryos using a method called preimplantation genetic screening (PGS) before they are implanted in the uterus to possibly increase their chances of having a successful pregnancy. One or more cells are removed from the embryo. The chromosomes inside the cells are then tested to identify normal or aneuploid embryo(s).

The investigators propose to evaluate a test called micro array analysis on the chromosomes of the first polar body. This method tests part of the egg that would normally be lost and may help us choose the embryo most likely to become a healthy baby.

DETAILED DESCRIPTION:
The polar body (PB) technique makes use of the 23 chromosomes contained in the first polar body, a part of the egg that is extruded at ovulation. Normally the first polar body disintegrates. However, it can be salvaged by polar body biopsy prior to this so that the chromosomes within can be analyzed. PB has three distinct advantages over conventional Fluorescent in-situ Hybridization (FISH) analysis. First, the polar body biopsy is performed on the day that the oocyte is retrieved (day 0) rather than day 3 so results are available earlier. Secondly, this methodology does not remove cells from the growing embryo. The polar body biopsy removes genetic material that would otherwise degrade. Finally, microarray analysis evaluates all 23 chromosomes while only 9-10 chromosomes can be studied with FISH analysis.

The investigators propose to perform microarray analysis in 50 IVF/ICSI (intracytoplasmic sperm injection) patients undergoing PGS.

Day 0 ICSI; PB* Day 1 Day 2 Day 3 Embryo biopsy with FISH or Microarray analysis Day 4 Day 5 Embryo transfer or embryo biopsy with Microarray analysis followed by Embryo Cryopreservation

Polar body biopsies will be frozen and later analyzed, The PB results will remain undisclosed until the end of the study period. PB results will not be used to guide treatment or clinical management. Embryos will be chosen or deselected for transfer solely based on the standard of care treatment aneuploidy screening analysis.

The three specific aims of the project are as follows:

* To determine the efficacy of PB biopsy and analysis by comparing the PB results to the Fluorescent in-situ Hybridization (FISH)/microarray results
* To evaluate the safety of PB by comparing the implantation , miscarriage, pregnancy, and delivery rates
* To determine the error rate of FISH analysis by analyzing the remaining cells in embryos determined to be abnormal by initial FISH/microarray analysis

ELIGIBILITY:
Inclusion Criteria:

1. Are undergoing IVF/Intracytoplasmic sperm injection(ICSI)
2. Are considering preimplantation genetic screening for aneuploidy
3. Are between ages 18 and 42 inclusive (female partner)

Exclusion Criteria:

1. Using sperm from a testicular source
2. Fewer than 10 oocytes retrieved
3. Fewer than 6 oocytes fertilized normally
4. Complete fertilization failure (no oocytes fertilize)

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of polar biopsy and preimplantation genetic analysis | 1 year
  To determine the efficacy of PB biopsy and analysis by comparing the PB results to the FISH/microarray results

SECONDARY OUTCOMES:
Safety of polar biopsy | 1 year
  To evaluate the safety of polar biopsy by comparing the implantation, miscarriage, pregnancy, and delivery rates

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Schattman, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Ronald O. Perelmand and Claudia Cohen Center for Reproductive Medicine, New York, New York, United States

REFERENCES:
- See also: Related Info — http://ivf.org